CLINICAL TRIAL: NCT02725957
Title: A Single Center, Single Ascending Dose, Double-Blind, Randomized, Placebo-Controlled Trial to Establish Safety and the Maximum Tolerated Dose of Intravenous Trehalose Solution in Healthy Subjects
Brief Title: A Study to Establish Safety and Maximum Tolerated Dose of IV Trehalose in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioblast Pharma Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: BB-TRE-101
Record Dates: First submitted 2016-03-15; First posted 2016-04-01 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer Subjects
Keywords: Bioblast
MeSH Terms: interventions — Trehalose; Infusions, Intravenous; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trehalose 9% (Experimental): Single dose administration of Trehalose 9% for IV infusion.
  Interventions: Drug: Trehalose for IV Infusion
- Saline 0.9% (Placebo Comparator): Single dose administration of 0.9% saline in the same volume and duration as Treatment Arm 1 (9% trehalose)
  Interventions: Drug: Saline 0.9% IV

INTERVENTIONS:
Drug: Trehalose for IV Infusion
  Arms: Trehalose 9%
Drug: Saline 0.9% IV
  Arms: Saline 0.9%

SUMMARY:
This will be a double-blind, randomized, placebo-controlled, single ascending dose study performed in healthy subjects.

The study will include up to four escalating dose cohorts with eight (8) subjects in each cohort.

In each cohort, eligible subjects will be randomized in a 3:1 ratio to receive single IV administration of 9% trehalose (Treatment Arm 1) or placebo (Treatment Arm 2).

All subjects, regardless of their treatment arm assignment, will undergo the same evaluations and will receive the study drug at the clinic. Each subject will continue to be followed for one week post dosing.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, single ascending dose study performed in healthy subjects.

The study will include up to four escalating dose cohorts with eight (8) subjects in each cohort.

In each cohort, eligible subjects will be randomized in a 3:1 ratio to receive single IV administration of 9% trehalose (Treatment Arm 1) or placebo (Treatment Arm 2).

All subjects, regardless of their treatment arm assignment, will undergo the same evaluations and will receive the study drug at the clinic. Each subject will continue to be followed for one week post dosing.

Cohorts 1 to 3 After all subjects in a given cohort complete their 1-week follow-up visit (Visit 4), a Safety Review Committee (SRC) will review the safety and PK data of that cohort. If no safety concerns are identified, and the exposure data supports a higher dose is acceptable, the SRC will approve continuation into the next cohort (dose level).

Cohort 4 Cohort 4 will be initiated based on review of the safety and exposure data from the first 3 cohorts by the SRC. This cohort will only be performed if there is a suggestion that exposure can be safely increased.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women between 18 and 55 years (inclusive) of age
2. Body Mass Index (BMI) 19 to 29.9 kg/m2 (inclusive) and weighing at least 55 kg.
3. Subjects in general good health in the opinion of the investigator
4. Blood pressure and heart rate within normal limits
5. Female subjects must have a negative serum pregnancy test during the Screening period (Day -28 to -1) and be willing and able to use a medically acceptable method of birth control or be postmenopausal.

Exclusion Criteria:

1. Diabetes mellitus type 1 or 2 or HbA1c > 5.6 % at Screening
2. History of significant medical disorder
3. Any clinically significant abnormality in safety laboratory tests during the Screening period (Day -28 to -1)
4. Known contraindication, hypersensitivity and/or allergy to trehalose
5. Any acute illness (e.g. acute infection) within 72 hours
6. Participation in another clinical trial with drugs received within 3 months prior to dosing
7. Positive serum pregnancy test determined during the Screening period or currently lactating women
8. ECG with clinically significant finding recorded during the Screening period
9. Positive HIV, Hepatitis B or Hepatitis C serology at Screening
10. Known history of alcohol or drug abuse in the past 5 years
11. Positive urinary drug screen determined during the Screening period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of escalating doses of intravenously administered trehalose (incidence of adverse events and serious adverse events, including clinically significant laboratory abnormalities) | Will be assessed during the entire study. At screening, at day -1 before drug administration, and day 1 of drug administration before, during and after drug administration, and at day 8 the follow up visit
  Safety will be assessed by the incidence of adverse events and serious adverse events, including clinically significant laboratory abnormalities.

SECONDARY OUTCOMES:
Maximum-tolerated dose (MTD) of trehalose administered intravenously (Averse events, vitals signs) | Will be assessed during the entire study. At screening, at day -1 before drug administration, and day 1 of drug administration before, during and after drug administration, and at day 8 the follow up visit
  The maximum-tolerated dose of trehalose will be assessed by evaluating the safety and tolerability of each of the escalating trehalose doses
Pharmacokinetics (PK) of plasma and urine trehalose | Will be assessed on the day of drug administration, before drug administration and up to 12hours following administration.
  To determine the pharmacokinetics (PK) of trehalose following administration of escalating doses of trehalose
Pharmacokinetics (PK) of serum and urine glucose | Will be assessed on the day of drug administration, before drug administration and up to 12hours following administration.
  To determine the pharmacokinetics (PK) of glucose following administration of escalating doses of trehalose

CONTACTS AND LOCATIONS:
Locations (1):
- PAREXEL Baltimore Early Phase Clinical Unit; Harbor Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided